CLINICAL TRIAL: NCT05381207
Title: Impact Of Montelukast On Allergic Rhinitis And Its Inflammatory Makers
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hadeer Ashraf Farouk, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Montelukast on A.R
Record Dates: First submitted 2022-05-08; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Allergic Rhinitis
Keywords: Montelukast; Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Montelukast (Active Comparator): Montelukast, 10 mg, oraly Local corticosteriod nasal spary
  Interventions: Drug: Montelukast Oral Tablet
- No drug (No Intervention): No drug taking , only local corticosteriod nasal spray

INTERVENTIONS:
Drug: Montelukast Oral Tablet — Subjects in group A (study) will be treated with Fluticasone Furoate nasal: (50 micrograms/spray) 100 micrograms (2 sprays) in each nostril twice daily plus oral montelukast (montelukast 10 mg, once a day) for 3 months. Subjects group B (control) will receive only topical steroids in an identical regimen
  Other Names: Fluticasone Furoate nasal spary
  Arms: Montelukast

SUMMARY:
To examine the efficacy of Montelukast as an adjunct to INCS in patients with allergic rhinitis.

DETAILED DESCRIPTION:
Allergic rhinitis (AR) is a non-infectious inflammatory disease occurring in nasal mucosa with nasal itching, nasal congestion, rhinorrhea, and sneezing as its main clinical symptoms, which are induced by immunoglobulin E-mediated chemical mediators with the participation of various immunologically competent cells and cytokines after allergen exposure. (1) According to statistics, AR affects 10% to 25% of the global population. (2).

AR could be investigated by skin prick test, A blood test to check for the immunoglobulin E (IgE) antibody, and Total blood eosinophil count. (3) Current guidelines suggest that Intranasal corticosteroids should be used as the first line of treatment (4).

Surgical care may be indicated for comorbid or complicating conditions such as chronic sinusitis and nasal polyps. (5) Many studies have proven that the abnormality of inflammatory factors such as(TNF-α, IL-6, and IL-12)are closely related to the pathogenesis of AR. (6)these inflammatory factors participate in the regulation of immune response through media leucocyte chemotaxis and activate, so elevate of levels of these 3 factors can reflect the aggravation of inflammatory markers in the patient with AR. (7) Montelukast is belonging to the leukotriene receptor antagonists with the effect of inhibiting the expression of cysteinyl leukotriene involved in the pathogen of AR. Thus, the inhibition of the inflammatory marker can effectively reduce airway inflammatory response, nasal mucosal edema, and inflammatory exudation etiologically [8].

ELIGIBILITY:
Inclusion Criteria:

Adult patients (aged 18 years and over) with AR. Clinical diagnosis of Allergic Rhinits Must be able to swallow tablets

Exclusion Criteria:

Bronchial Asthma patients. Patients already on Antihistamine combined treatment Patients who are allergic to this medication Advanced liver or kidney diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Nasal symptoms | 3 monthes
  Participants will be asked to score five Sino-nasal symptoms (nasal congestion/obstruction, anterior rhinorrhea, posterior rhinorrhea, loss of smell, and facial pain) from 0 to 4.
  This score will be assessed at the screening and follow-up visits at 12 weeks. The total five-symptom score (T5SS) was obtained with the sum of the individual symptoms (0-20).
laboratory findings | 3 months
  Evaluation of inflammatory markers levels (TNF-α, IL-6, IL-12) in inpatient blood At 0 point premedication (pre-medication) At 1 point post medication after 12 weeks (3 months)
Quality of life symptoms | 3 monthes
  Subjects will complete a validated questionnaire related to the general quality of life in patients with allergic rhinitis; this questionnaire records patients' symptoms The patients receive a rhino-conjunctivitis quality of life questionnaire. This questionnaire records domains like patient activities, sleep, ......and emotional problems on an 0-x ordinal scale.

IPD SHARING:
Plan to Share IPD: Undecided